CLINICAL TRIAL: NCT02900768
Title: Evaluating Effects on Quality of Life of a Partially Supervised Exercise Program Following Allogeneic Stem Cell Transplantation
Brief Title: Effects of Exercise on Allogeneic Stem Cell Transplant
Acronym: Ex-BMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Raewyn Broady (Other)
Responsible Party: Sponsor-Investigator, Raewyn Broady, Clinical Associate Professor, University of British Columbia
Organization: University of British Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H16-00112
Record Dates: First submitted 2016-08-14; First posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Hematological Malignancy
Keywords: Bone Marrow Transplantation; Exercise; Rehabilitation; Cancer
MeSH Terms: conditions — Hematologic Neoplasms; Motor Activity; Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise Group (Experimental): Patients in the intervention group will receive supervised and unsupervised exercise program after their bone marrow transplant.
  Interventions: Behavioral: Exercise
- Control Group (No Intervention): Patient will receive standard of care within the hospital as an inpatient and outpatient after their bone marrow transplant.

INTERVENTIONS:
Behavioral: Exercise — Combination of resistance and aerobic exercises for 100 days.
  Arms: Exercise Group

SUMMARY:
Although allogeneic haematopoietic stem cell transplant (AlloHSCT) is a curative treatment option for malignant hematological diseases, it is also associated with significant morbidity such as graft versus host disease, infections, and immune complications. Moreover, long-term survivors are likely to have reduced physical performance and functioning due to deconditioning, sarcopenia, and bone loss, and particularly high levels of fatigue and psycho-social stress, all of which negatively impact patients' quality of life.

Purpose: To conduct a randomized controlled, single site trial investigating whether a partially supervised exercise intervention in the first 100 days post alloHSCT patients will result in improved quality of life at Day 100 post-transplant compared to standard of care treatment. Secondary objectives will investigate the effect of an exercise intervention on muscle strength, cardiorespiratory fitness, mobility, bone mineral density, body composition, exercise, and immunological/inflammatory biomarkers compared to standard of care.

Procedure: 120 patients receiving alloHSCT will be baseline tested, and then randomized into an Exercise Intervention Group or Standard of Care Control Group.

DETAILED DESCRIPTION:
This is a randomized non-blinded single centre prospective clinical trial designed to evaluate the efficacy and safety of a partially-supervised progressive exercise intervention among patients undergoing alloHSCT compared to a self-directed exercise program. Approximately 120 patients will be enrolled. Following completion of all baseline data collection, participants will be randomized 1:1 to the intervention group or the control group.

Patients in the intervention group will receive an exercise manual with background information, descriptions for different resistance and aerobic exercises, and instructions for tailoring the intensity of exercise. All patients will receive Therabands™ for resistance exercises and have access to a stationary bicycle for aerobic exercises with practical introduction by an exercise specialist. The partially supervised intervention is a progressive program with a goal of three aerobic and two resistance exercise sessions per week.

Aerobic exercise will consist of 10-30 minutes of bicycling using a stationary bike (supervised or unsupervised) or brisk walking, following the Borg Scale of Rate of Perceived Exertion (RPE). Resistance exercise will include exercise for the upper and lower extremities with Therabands™. Exercise will be adapted based on the participant's clinical status for safety and ability to perform exercises. At the weekly supervised session, the exercise specialist will provide adequate progression of exercises, and review adherence to the intervention and provide support for questions and overcoming identified barriers to adherence.

Participants assigned to the control group will receive our current standard of care. They will be reviewed by the ward physiotherapist on admission to hospital and encouraged to maintain physical activity by walking around the inpatient unit during their inpatient hospitalization. As per standard of care, the physiotherapist will be available on an as needed basis in both the inpatient and outpatient settings.

Timely assessments of outcome measures outlined in the "Outcome Measures" section will be conducted for both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing allogeneic stem cell transplantation (including related, unrelated, cord blood or haploidentical allogeneic transplant) for any indication through the Leukemia/BMT Program of British Columbia.
2. Age greater than or equal to 18 years.
3. Able to provide written informed consent.

Exclusion Criteria:

1. Severe cardiac disease including symptomatic congestive heart failure (New York Heart Association Class III or IV), unstable angina pectoris, or an unstable cardiac arrhythmia.
2. Orthopedic illness which limits ability to conduct aerobic exercise (walking or biking).
3. Not meeting eligibility criteria to proceed with allogeneic stem cell transplantation as per the Leukemia/BMT Program of BC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-09; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life | Baseline, Day 100 post-transplant
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire.
  To investigate if a partially supervised exercise intervention in alloHSCT patients will result in differences in quality of life at Day 100 post transplant compared to the standard of care control group.

SECONDARY OUTCOMES:
Changes in Quality of Life | Baseline, Hospital Discharge (approximately +30 days post-transplant), Day 60, 100, 365, and 730 post-transplant
  EuroQol (EQ)-5 Dimensions (5D) -3 Level (3L) Questionnaire.
Changes in Grip Strength | Baseline, Hospital Discharge (approximately +30 days post-transplant), Day 60, 100, 365, and 730 post-transplant
  Using a handheld dynamometer, measured in kg.
Changes in 30-Second Chair Stand | Baseline, Hospital Discharge (approximately +30 days post-transplant), Day 60, 100, 365, and 730 post-transplant
  Number of chair stands one can perform in 30 seconds.
Changes in 6-Minute Walk Test | Baseline, Hospital Discharge (approximately +30 days post-transplant), Day 60, 100, 365, and 730 post-transplant
  Distance (meters) someone can walk in 6 minutes between two cones separated by 30 meters.
Changes in Timed Up and Go | Baseline, Hospital Discharge (approximately +30 days post-transplant), Day 60, 100, 365, and 730 post-transplant
  Time taken for someone to stand up from a chair, walk 3 meters, turn around, walk back to the chair, and sit sound.
Changes in Exercise Capacity | Baseline, Day 100, 365, and 730 post-transplant
  Exercise Treadmill Test via Bruce or Modified Bruce Protocol. METs and estimated peak oxygen uptake (VO2) will be determined.
Changes in Cardiopulmonary Function | Baseline, Day 100, 365, and 730 post-transplant
  Left ventricular ejection fraction vs radionuclide ventriculography (MUGA) or echocardiography.
Changes in Physical Activity Levels - Accelerometry | Baseline, Hospital Discharge (approximately +30 days post-transplant), Day 60, 100, 365, and 730 post-transplant
  Accelerometry counts converted minutes/week of moderate-to-vigorous activity and sedentary activity and METS. Godin Leisure-Time Exercise Questionnaire.
Changes in Physical Activity Levels - Questionnaire | Baseline, Hospital Discharge (approximately +30 days post-transplant), Day 60, 100, 365, and 730 post-transplant
  Godin Leisure-Time Exercise Questionnaire. Total leisure activity score is calculated.
Changes in Body Composition Analysis | Baseline, Hospital Discharge (approximately +30 days post-transplant), Day 60, 100, 365, and 730 post-transplant
  Height (cm), weight (m), and waist/hip circumference (cm) will be measured.
Changes in Bone Mineral Density Analysis | Baseline, Day 100, 365, and 730 post transplant
  Bone mineral density testing will be performed using a Dual-Energy X-Ray Absorptiometry (DXA).
Changes in Immune Biomarkers | Baseline, Day 100, 365, and 730 post-transplant
  A collective blood test will be done to determine the composition of white blood cells (total, lymphocytes, and subsets of T-Lymphocytes).

CONTACTS AND LOCATIONS:
Overall Officials: Alina Gerrie, MD, FRCPC, Principal Investigator — British Columbia Cancer Agency; Raewyn Broady, MBChB, FRCPC, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided